CLINICAL TRIAL: NCT06745362
Title: Weight Reduction With the Low-Insulin-Method - Self Monitoring of Breath Acetone
Acronym: WeR-LIM-SMBA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20241217
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Overweight and Obese Volunteers
Keywords: lifestyle intervention; weight reduction; ketosis
MeSH Terms: conditions — Overweight; Weight Loss; Ketosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): lifestyle intervention including information about ketosis level
  Interventions: Other: self-monitoring of breath acetone; Other: lifestyle-intervention via LIM-App
- control group (Active Comparator): lifestyle intervention without information about ketosis level
  Interventions: Other: lifestyle-intervention via LIM-App

INTERVENTIONS:
Other: self-monitoring of breath acetone — Participants perform self-monitoring of braeth acetone in order to get information about their ketosis state.
  Arms: Intervention group
Other: lifestyle-intervention via LIM-App — Participants are offered a lifestyle intervention via LIM-App.

SUMMARY:
The goal of this clinical trial is to learn if lifestyle intervention with information about ketosis state supports weight reduction in overweight adults.

Researchers will compare an App-based lifestyle intervention with self-monitoring of breath acetone vs. lifestyle intervention alone.

Participants will:

Get a lifestyle intervention via the LIM-App for 12 months. Report body weight.

DETAILED DESCRIPTION:
Background: Overweight and obesity are an increasing problem. Therefore, the Low-Insulin-Method was developed to support overweight and obese people in weight loss.

Method: In a randomized controlled clinical trial, the effect of the lifestyle intervention program 'Low-Insulin-Method', delivered by the Low-Insulin-App including low-carb diet, physical activity, self monitoring of weight, and self-monitoring of breath acetone (SMBA) is examined compared to a control group without information about ketosis level. Weight change will be compared after 3 and 12 months.

Objective: The aim is to develop a training and counseling program for overweight or obese individuals with diabetes risk or type 2 diabetes, which can be used both for primary and for tertiary prevention of overweight-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > 25kg/m2

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
body weight | 3 months
  body weight in kg

SECONDARY OUTCOMES:
body weight | 12 months
  body weight in kg

CONTACTS AND LOCATIONS:
Locations (1):
- West German Center of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No
upon request